CLINICAL TRIAL: NCT01350869
Title: Evaluation of Effectiveness and Safety of Everolimus-Eluting Stents in Routine Clinical Practice
Brief Title: Evaluation of Everolimus-Eluting Stents (The K-XIENCE Registry)
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: 2009-0588
Record Dates: First submitted 2011-04-22; First posted 2011-05-10 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Xience stent: Real world patients treated with XIENCE stents
  Interventions: Device: Xience

INTERVENTIONS:
Device: Xience — Patients with Xience

SUMMARY:
The objective of this study is to evaluate effectiveness and safety of everolimus-eluting stents (XIENCE, Abbott) in the "real world" daily practice as compared with first-generation drug-eluting stents (sirolimus-eluting stents).

DETAILED DESCRIPTION:
This study is a non-randomized, open-label registry to compare the efficacy and safety of everolimus-eluting stents versus sirolimus-eluting stents in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients received XIENCE stents
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Patients with a mixture of other DESs
* Terminal illness with life expectancy <1 year.
* Patients with cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will be conducted at 33 centers in Korea. Data will be collected on approximately 3,000 subjects treated with XIENCE stents.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Composite of death, nonfatal myocardial infarction (MI), and Target Vessel Revascularization (TVR) | at 12 months after PCI
  composite of death, nonfatal myocardial infarction (MI), or ischemic driven Target Vessel Revascularization (TVR). Individual events are to be assessed as secondary.

SECONDARY OUTCOMES:
All Death | 1month ,6 month and 12 months,2year,3year,4 year and 5year
  1month ,6 month and 12 months,2year,3year,4 year and 5year
Cardiac death | 1month ,6 month and 12 months,2year,3year,4 year and 5year
  1month ,6 month and 12 months,2year,3year,4 year and 5year
MI | 1month ,6 month and 12 months,2year,3year,4 year and 5year
  1month ,6 month and 12 months,2year,3year,4 year and 5year
Composite of death or MI | 1month ,6 month and 12 months,2year,3year,4 year and 5year
  1month ,6 month and 12 months,2year,3year,4 year and 5year
Composite of cardiac death or MI | 1month ,6 month and 12 months,2year,3year,4 year and 5year
  1month ,6 month and 12 months,2year,3year,4 year and 5year
TVR | 1month ,6 month and 12 months,2year,3year,4 year and 5year
  1month ,6 month and 12 months,2year,3year,4 year and 5year
Target-lesion revascularization (TLR) | 1month ,6 month and 12 months,2year,3year,4 year and 5year
  1month ,6 month and 12 months,2year,3year,4 year and 5year
Stent thrombosis (ARC criteria) | 1month ,6 month and 12 months,2year,3year,4 year and 5year
  1month ,6 month and 12 months,2year,3year,4 year and 5year
Procedural success | at discharge
  defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, Seoul, South Korea